CLINICAL TRIAL: NCT02207166
Title: Identify Possible Errors on Home Use Blood Pressure Monitors by Usability Reasoning (IPEOHUBPMBUR)
Brief Title: Identify Possible Errors on Home Use Blood Pressure Monitors by Usability Reasoning
Acronym: IPEOHUBPMBUR
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201406066RINB
Record Dates: First submitted 2014-07-27; First posted 2014-08-04 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Hypertension
Keywords: hypertension; device; errors; human factor engineering; usability engineering
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- user group: volunteers who are willing to receive 40 minutes video monitoring and questionnaires while operation a electronic blood pressure measuring machines.

SUMMARY:
Medical devices are designed and manufactured by subjective design process that was only based on engineers' direct concepts to essential principles sets for the device. A home user may not easily use or operate the piece of medical device through the interfacing components as the designer's expected such as the meaning when pushing a button or switching a knob, even the required procedure needed when a certain display shown to fulfill some knowledge dependent judgment. In addition, the incompatible interfacing designed communication between a user and the device may cause possible errors that may trigger further negative consequences during the use of the device to a innocent home user.

The aim of this research is to closely understand the consequent results of human factor engineering or usability engineering practices of various types or models of marketed home-use blood pressure monitors (BPM) in real use.

DETAILED DESCRIPTION:
The aim of this research is to closely understand the consequent results of human factor engineering or usability engineering practices of various types or models of marketed home-use blood pressure monitors (BPM) in real use. Participants of the intended user population interact with marketed BPMs in research to assess ease of learning, ease of use, effectiveness and efficiency of use, memorability, safety, and/or user appeal among the many possible attributes of interest. With these understanding and analysis of human factors engineering / usability engineering (HFE/UE) practiced status, it can help manufacturers to capture the required and diversified HFE/UE essences with the minimum or limited professional technical resources in hand some more efficiently.

ELIGIBILITY:
Inclusion Criteria:

* age between 20-75 years
* capable of operating the blood pressure measure machine provided by the study
* willing to operate the provided device and accept video taping from shoulder and below
* willing to fill the study questionnaire and to provide feedback after use of the device

Exclusion Criteria:

* vulnerable population (including pregnant woman, disabled, etc)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who are able to operate general healthcare devices (eg thermometer, electronic blood pressure measures)
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Total steps of incorrect operations | During the 40-60 mins osbervation period
  Possible errors may cause negative outcomes to a home-user when he/she uses the BPM. The principal concept of "usability" is that a good usability designed BPM is easy to operate it as the device designer expected a home-user to perform in real use.

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan